CLINICAL TRIAL: NCT05888740
Title: A Prospective, Non-significant Risk, Feasibility Study to Evaluate Serial Applications of VibratoSleeve Therapy to Acutely Increase the Perfusion in Peripheral Arterial Disease (PAD) Subjects 65 Years of Age and Older
Brief Title: Feasibility Study to Evaluate Therapeutic Ultrasound (TUS) to Acutely Increase the Perfusion in Peripheral Arterial Disease (PAD)
Acronym: Waltz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrato Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022-01
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Therapeutic Ultrasound (TUS); Peripheral Artery Disease (PAD); Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, open-label, feasibility acute phase study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- TUS Therapy (Experimental): These subjects will undergo treatments with the Vibrato Sleeve TUS device.
  Interventions: Device: VibratoSleeve Therapeutic Ultrasound Device

INTERVENTIONS:
Device: VibratoSleeve Therapeutic Ultrasound Device — The VibratoSleeve is compromised of a 16-transducer array that is mounted within a wrap that conforms to the posterior calf

SUMMARY:
This study is evaluating whether a therapeutic ultrasound device can improve symptoms in the leg of peripheral arterial disease (PAD) patients 65 years of age and over.

DETAILED DESCRIPTION:
The VibratoSleeve TUS will be used on to assess its acute vasodilatory and perfusion effects in subjects with early stage PAD. Each subject will receive TUS treatment multiple sessions. All post- treatment acute assessments will take place immediately following each day's treatment and no follow-up assessments will be required in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65
2. Diagnosis of PAD.
3. Claudication symptoms in Rutherford class 1,2, or 3 as determined by the investigator.

Exclusion Criteria:

1. Prior stenting in posterior tibial artery.
2. Re-vascularization procedure within 30 days prior to enrollment in the study.
3. Ulcers, cellulitis, or skin breakdown in treatment areas (posterior calf).
4. History or diagnosis of severe chronic venous insufficiency.
5. Acute limb ischemia within 30 days prior to treatment.
6. History or diagnosis of deep venous thrombosis below the knee in treatment leg.
7. Any conditions that, in the opinion of the investigator, may render the subject unable to complete the study or lead to difficulties for subject compliance with study requirements, or could confound study data.
8. Subject's enrollment in another investigational study that has not completed the required primary endpoint follow-up period.

stenting in posterior tibial artery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular & Interventional Specialists of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nazer B, Ghahghaie F, Kashima R, Khokhlova T, Perez C, Crum L, Matula T, Hata A. Therapeutic Ultrasound Promotes Reperfusion and Angiogenesis in a Rat Model of Peripheral Arterial Disease. Circ J. 2015;79(9):2043-9. doi: 10.1253/circj.CJ-15-0366. Epub 2015 Jun 9. PMID 26062950

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TUS Therapy
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TUS Therapy
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Acute Flow Rate Difference During TUS Treatment Sessions
Description: Percent change in perfusion measured by FlowMet calculated between baseline and after final treatment.
Time Frame: Baseline to end of treatment, an average of 1 month
Measure: Mean (Standard Deviation); unit: Percent change (%)
Arm/Group | TUS Therapy
Number analyzed (Participants) | 12
Percent change (%) | 27.3 (50.8)

2. Primary Outcome: Tissue Oxygen Saturation (StO2)
Description: Calculate changes in tissue oxygen saturation (StO2) measured non-invasively by Clarifi spatial frequency domain imaging system, compared from baseline to during and immediately post-treatment.
Time Frame: Through study completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: StO2%
Arm/Group | TUS Therapy
Number analyzed (Participants) | 12
StO2% | 1.0 (8.4)

3. Primary Outcome: Ankle Brachial Index (ABI)
Description: ABI is ratio that compares blood pressure in the arm to blood pressure in the ankle. It is a measurement of the extent of peripheral arterial disease.
Time Frame: Baseline to end of treatment, an average of 1 month
Measure: Mean (Standard Deviation); unit: Index (Ratio)
Arm/Group | TUS Therapy
Number analyzed (Participants) | 12
Index (Ratio) | 0.0 (0.12)

4. Secondary Outcome: Incidence of Device and Procedure-related Adverse Events
Description: Number of adverse events related to the VibratoSleeve device or study procedure occurring throughout the duration of the study.
Time Frame: Through study completion, an average of 1 month
Measure: Number; unit: Events
Arm/Group | TUS Therapy
Number analyzed (Participants) | 12
Events | 0

ADVERSE EVENTS:
Time Frame: Safety surveillance and reporting starts when subject receives therapy with the VibratoSleeve until the end of the final treatment visit. All treatment visits were completed within an average of 1 month per patient.
Description: Although unlikely due to the nature of the device, the following adverse events were reported for each subject through the final treatment visit:
  All device-related adverse events and events for which the relationship to the VibratoSleeve is unknown
  All SAEs Unchanged, chronic, non-worsening or pre-existing conditions are not AEs and should not be reported. Planned hospitalization for a pre-existing condition is not considered a serious adverse event.
Arm/Group | TUS Therapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish data obtained from the Study provided that the Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for written approval, for which approval shall not be unreasonably denied. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor (including trade secrets but not including Results) from the proposed publication or presentation.

DOCUMENTS (1):
  • Study Protocol (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT05888740/Prot_001.pdf